CLINICAL TRIAL: NCT04574817
Title: A Single-arm, Open-lable, Multicenter, Phase II Clinical Study of HX008 in Subjects With Anaplastic Thyroid Cancer
Brief Title: Study of HX008 for the Treatment of Anaplastic Thyroid Cancer (ATC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taizhou Hanzhong biomedical co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX008-II-ATC-01
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Anaplastic Thyroid Cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HX008 (Experimental): Participants will receive HX008 200 mg intravenous (IV) every 3 weeks (Q3W)
  Interventions: Drug: HX008

INTERVENTIONS:
Drug: HX008 — 200 mg administered as IV infusion on Day 1 of each 21-day cycle.

SUMMARY:
There are currently no target therapies approved for treatment of anaplastic thyroid cancer (ATC), leading to a clear need for improving therapy for ATC. This is a single-arm, multicenter study to evaluate the efficacy and safety of HX008 injection in patients with metastatic or locally advanced anaplastic thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Age ≥ 18 years old, male or female.
* Subjects must have histological diagnosis of inoperative IVB or IVC stage anaplastic thyroid cancer.
* Prior neoadjuvant, adjuvant or palliative chemotherapy for ATC is allowed, there is no limit to the number of prior lines of treatment a patient has received.
* Have measurable disease based on RECIST 1.1.
* Willing to provide tissue for PD-L1 biomarker analysis.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Score.
* Life expectancy ≥ 3 months.
* Has adequate organ function as defined in the protocol.
* Female subject of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of study treatment.
* Male and female participants should agree to use an adequate method of contraception during the experiment and 6 months after the last administration of the test drugs.

Exclusion Criteria:

* Subjects who are suitable or intent to receive local treatment.
* Differentiated thyroid cancer (DTC) or medullary thyroid cancer (MTC). ATC arising out of DTC is allowed, as long as the measurable disease is clinically consistent with ATC i.e., rapidly progressive and/or 18F fluorodeoxyglucose (FDG)-avid.
* Subjects diagnosed with any other malignancy within 3 years prior to the first dose of HX008, except for malignancies with a low risk of metastasis and death (5-year survival rate > 90%), such as basal cell or squamous cell skin cancer or carcinoma in situ of the cervix and other carcinomas in situ.
* Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to the first dose of trial treatment or who has not recovered (≤ Grade 1 or at Baseline) from AEs due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, radiation therapy or targeted small molecular therapy within 2 weeks prior to the first dose of trial treatment or who has not recovered (≤ Grade 1 or at Baseline) from AEs due to a previously administrated agent.
* Has had prior herbal medicine within 1 week prior to the first dose of trial treatment.
* Has received prior therapy with an anti-PD-1, or anti-PD-L1, or anti-CTLA-4 agents.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in past 2 years.
* Has received a major surgery within 4 weeks prior to the first dose of trial treatment.
* Has received system treatment with corticosteroids (dose >10mg/day prednison or other therapeutic hormones) within 2 weeks prior to the first dose of trial treatment.
* Has a history of interstitial lung disease.
* Has uncontrolled cardiovascular disease, including but not limited to: 1) heart failure greater than New York Heart Association (NYHA) class II; 2) unstable angina pectoris; 3) has myocardial infarction within 1 year; 4) supraventricular or ventricular arrhythmias with clinical significance.
* Has uncontrolled systemic disease, such as diabetes or hypertension.
* Has a history of active tuberculosis.
* Has a history of testing positive for human immunodeficiency virus (HIV), or known acquired immunodeficiency syndrome (AIDS), or stem cell transplantation or organ transplantation.
* Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
* Has untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 500 IU/ mL or active hepatitis C virus (HCV). Subjects with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA < 10^3 copies/ml or <500 IU/ mL) , and cured hepatitis C can be enrolled. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
* Has a history of severe allergic reaction to any other monoclonal antibodies.
* Has active infections requiring systemic treatment within 2 weeks prior to the first dose of trial treatment.
* Has participated in other anticancer drug clinical trials within 4 weeks.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-12-28 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 30 months
  Percentage of subjects achieving complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to approximately 30 months
  DCR was defined as the percentage of participants who have a CR or a PR or a stable disease (SD)
Duration of Response (DOR) | Up to approximately 30 months
  DOR was defined as the time from the first documented evidence of a response of CR or PR to the first documented disease progression or death due to any cause, whichever occurs first.
Progression-free Survival (PFS) | Up to approximately 30 months
  PFS was defined as the time from the date of beginning of HX008 administration to the first documented disease progression or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 30 months
  OS was defined as the time from the date of beginning of HX008 administration until date of death from any cause.
Adverse Effect (AE) | Up to approximately 30 months
  Adverse events associated with HX008

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China